CLINICAL TRIAL: NCT05737069
Title: A Randomized, Open-label, Single-center, Single-dose, Two Treatment, Two-sequence, Two-period, Two-cohort, Two-way Crossover Bioequivalence Study of Two Ibuprofen Arginine Granules 400 mg Formulations Under Fasting and Fed Conditions in Chinese Healthy Adult Subjects
Brief Title: A Bioequivalence Study of Two Ibuprofen Arginine Granules 400 mg Formulations Under Fasting and Fed Conditions in Chinese Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 218552
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — ibuprofen arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen arginine granules 400 mg (Experimental): Participants will be randomly assigned as per cross-over design to receive one sachet of Ibuprofen arginine granules 400 mg (test product) on day 1 of period 1 and will receive one sachet of Ibuprofen arginine granules 400 mg (Spedifen) (reference product) on day 1 of period 2 with at least 2 days washout period. Participants will be instructed to consume the product orally by dissolving it in 240 mL of warm water.
  Interventions: Drug: Ibuprofen arginine granules 400 mg; Drug: Ibuprofen arginine granules 400 mg (Spedifen)
- Ibuprofen arginine granules 400 mg (Spedifen) (Active Comparator): Participants will be randomly assigned as per cross-over design to receive one sachet of Ibuprofen arginine granules 400 mg (Spedifen) (reference product) on day 1 of period 1 and will receive one sachet of Ibuprofen arginine granules 400 mg (test product) on day 1 of period 2 with at least 2 days washout period. Participants will be instructed to consume the product orally by dissolving it in 240 mL of warm water.
  Interventions: Drug: Ibuprofen arginine granules 400 mg; Drug: Ibuprofen arginine granules 400 mg (Spedifen)

INTERVENTIONS:
Drug: Ibuprofen arginine granules 400 mg — Experimental- Ibuprofen arginine granules 400 mg, one sachet administration containing 400 mg ibuprofen granules.
Drug: Ibuprofen arginine granules 400 mg (Spedifen) — Marketed drug- Ibuprofen arginine granules 400 mg (Spedifen), one sachet administration containing 400 mg ibuprofen granules.

SUMMARY:
The primary purpose of this study is to demonstrate the bioequivalence of two ibuprofen arginine granules 400 milligram (mg) formulations under fasting and fed conditions in Chinese healthy adult participants. The secondary purpose of this study is to assess the pharmacokinetic and safety profile of the test and reference preparations.

DETAILED DESCRIPTION:
The bioequivalence study adopts a single-center, randomized, open-label, single-dose, two-treatment, two-sequence, two-period, two-cohort, two-way crossover design with at least 2-day washout period, under both fasting and fed conditions in Chinese healthy adult participants. It will be planned to enroll approximately 84 participants out of which the first 34 participants for the fasted cohort and the subsequent 50 participants for the fed cohort receiving ibuprofen arginine granules 400 mg. Participants will be randomly assigned to either one of the 2 treatment (Test or Reference product) sequences in a 1:1 ratio within fasted cohort and fed cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants provision of a signed and dated informed consent and/or assent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participants who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, study restrictions, lifestyle considerations and other study procedures.
* Healthy Participants, which is defined as in general good physical health, as judged by the investigator and no clinically significant relevant abnormalities identified by a detailed medical history, full physical examination, including vital signs, 12-lead electrocardiogram (ECG) and laboratory tests.
* A Participants with a Body Mass Index (BMI) of 19-26 kilogram per meter square (kg/m^2) (including 19, excluding 26) [BMI equal to (=) weight (Kilogram [kg])/height^2 (m^2)]; and a total body weight more than or equal to >= 50 kilogram (kg) for males, and >= 45 kg for females, at screening.
* Participants with one negative polymerase chain reaction (PCR) or antigen test (on Day-1) for active Coronavirus disease 2019 (COVID-19).
* Participants of childbearing potential and are sexually active and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. Female participant who are not of childbearing potential must meet requirements in the Contraception section of protocol.

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity or photosensitivity to the investigational products (or closely related compounds) or any of their stated ingredients.
* Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the investigator's opinion may pose a risk to the candidate.
* Diagnosis of long QT syndrome or QTcF > 450 millisecond (msec) at screening.
* Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 millimeters of mercury (mmHg), diastolic blood pressure lower than 60 or over 90 mmHg, or pulse rate less than 50 or over 100 beats per minute [bpm]).
* Use of any medication (including over-the-counter medications and Chinese herbal and traditional remedies) within 2 weeks before first scheduled study drug administration or within less than 10 times the elimination half-life of the concomitant medication (whichever is longer) or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:

  1. systemic contraceptives and hormone replacement therapy, as long as female participant is on stable treatment for at least 3 months before first scheduled study drug administration and continues treatment throughout the study.
  2. occasional use of acetaminophen (up to 2 grams [g] in 24 hours).
* Participants has a history of drug abuse or has positive urine drug abuse screening at screening or on Day-1.
* Participants reported regular consumption of > 5 cups (1 cup approximately 250 milliliters [mL]) of coffee or tea per day (or equivalent consumption of >= 500 mg caffeine per day using other products). Or consuming any beverages or food containing caffeine, such as coffee, tea, coke, chocolate, etc., within 48 hours prior to screening.
* Smoking or history of regular use of tobacco- or nicotine-containing products (for example nicotine patch, electronic cigarette) within 6 months prior to screening. Or a participant who is unwilling to abstain from tobacco or nicotine containing product use during the study.
* Evidence, as reported by an alcohol breath testing, for current alcohol abuse or reports a regular average alcohol consumption exceeding 18 g (women) or 35 g (men) of pure alcohol per day, that is (i.e.) 1 drink/day for women or 2 drinks/day for men [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months prior to screening.
* Participation in other clinical trials involving investigational drug(s) within 90 days prior to screening.
* Those who have blood donation (including component donation) or blood loss >= 400 mL within 3 months before the study or have blood transfusion; those who have blood donation (including component donation) or blood loss >= 200 mL within 1 month before the study (except female physiological blood loss).
* Acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study. Or any condition not identified in the protocol that in the opinion of the investigator would confound the evaluation and interpretation of the study data or may put the participant at risk.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
* Participation with known COVID-19 positive contacts in the past 14 days.
* Participation with signs or symptoms highly suggestive of COVID-19 (including not limited to fever, cough, chills, new loss of taste or smell, etc.) that also align with the clinical judgement of the investigator, within 14 days of inpatient admission as defined by World Health Organization (WHO) or local guidance.
* Any vaccination, including COVID-19 vaccine, within 14 days prior to the first dose of investigational products.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance but not limited to any of the following:

  1. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, e.g., appendectomy and herniorrhaphy).
  2. History of inflammatory bowel disease.
  3. History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of estimated glomerular filtration rate (eGFR) less than (<) 90 mL/min/1.73m^2 or the presence of clinically significant abnormal urinary constituents (e.g., albuminuria).
  4. History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found:

     1. Aspartate aminotransferase (AST) (>= 1.2 upper limit of normal [ULN]), alanine transaminase (ALT) (>= 1.2 ULN),
     2. Gamma-glutamyl transferase (GGT) (>= 1.2 ULN), alkaline phosphatase (ALP) (>= 1.2 ULN),
     3. Bilirubin (>= 1.5 ULN) or creatine kinase (CK) (>= 3 ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the investigator.
  5. Evidence of urinary obstruction or difficulty in voiding at screening.
  6. History or clinical evidence at screening of pancreatic injury or pancreatitis.
* Pregnant or lactating women, or participant intending to become pregnant over the duration of the study.
* Positive results (or out of normal range) any of the virology tests for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody or syphilis.
* Participants reports consumption of any drug metabolizing enzyme (for example (e.g.), CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (e.g., broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort etc.) within 2 weeks prior to screening until admission to the unit.
* Performance of strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission.
* Those who are not suitable for participation in this study as determined by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Xu, Master, Principal Investigator — Clinical Pharmacological Research Center
Locations (1):
- Clinical Pharmacological Research Center, Wenjiang, Chengdu, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in China.
Pre-assignment Details: A total of 235 participants were screened of which 34 participants were enrolled in fasted cohort and 50 participants were enrolled in fed cohort. Participants were randomized in 1:1 ratio within each cohort (fasted and fed) to receive either one of the 2 treatment sequence: Test (T) product followed by Reference (R) product (TR) or Reference product followed by Test product (RT) as per cross-over design.
Groups:
- Fasted Cohort: Test Product-Reference Product (TR): Participants received one sachet of ibuprofen arginine granules 400 milligrams (mg) (test product), orally, once on Day 1 of Period 1 under fasting conditions followed by one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 2 under fasting conditions. Participants were instructed to take the study product after an overnight fast of at least 10 hours by dissolving it in 240 milliliters (mL) of warm water. There was a wash-out period of at least two days between the administration of each product.
- Fasted Cohort: Reference Product-Test Product (RT): Participants received one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 1 under fasting conditions followed by one sachet of ibuprofen arginine granules 400 mg (test product), orally, once on Day 1 of Period 2 under fasting conditions. Participants were instructed to take the study product after an overnight fast of at least 10 hours by dissolving it in 240 mL of warm water. There was a wash-out period of at least two days between administration of each product.
- Fed Cohort: Test Product-Reference Product (TR): Participants received one sachet of ibuprofen arginine granules 400 mg (test product), orally, once on Day 1 of Period 1 under fed conditions followed by one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 2 under fed conditions. Participants were instructed to take the study product after a high-fat/high-calorie meal by dissolving it in 240 mL of warm water. There was a wash-out period of at least two days between the administration of each product.
- Fed Cohort: Reference Product-Test Product (RT): Participants received one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 1 under fed conditions followed by one sachet of ibuprofen arginine granules 400 mg (test product), orally, once on Day 1 of Period 2 under fed conditions. Participants were instructed to take the study product after a high-fat/high-calorie meal by dissolving it in 240 mL of warm water. There was a wash-out period of at least two days between administration of each product.
Period: Period 1 (2 Days)
Arm/Group | Fasted Cohort: Test Product-Reference Product (TR) | Fasted Cohort: Reference Product-Test Product (RT) | Fed Cohort: Test Product-Reference Product (TR) | Fed Cohort: Reference Product-Test Product (RT)
Started | 17 | 17 | 25 | 25
Completed | 17 | 17 | 25 | 25
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (2 Days)
Arm/Group | Fasted Cohort: Test Product-Reference Product (TR) | Fasted Cohort: Reference Product-Test Product (RT) | Fed Cohort: Test Product-Reference Product (TR) | Fed Cohort: Reference Product-Test Product (RT)
Started | 17 | 17 | 25 | 25
Completed | 17 | 17 | 25 | 25
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (2 Days)
Arm/Group | Fasted Cohort: Test Product-Reference Product (TR) | Fasted Cohort: Reference Product-Test Product (RT) | Fed Cohort: Test Product-Reference Product (TR) | Fed Cohort: Reference Product-Test Product (RT)
Started | 17 | 17 | 25 | 25
Completed | 17 | 17 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population included all randomized participants.
Groups:
- Fasted Cohort: Test Product-Reference Product (TR): Participants received one sachet of ibuprofen arginine granules 400 mg (test product), orally, once on Day 1 of Period 1 under fasting conditions followed by one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 2 under fasting conditions. Participants were instructed to take the study product after an overnight fast of at least 10 hours by dissolving it in 240 mL of warm water. There was a wash-out period of at least two days between the administration of each product.
- Total: Total of all reporting groups
Arm/Group | Fasted Cohort: Test Product-Reference Product (TR) | Fasted Cohort: Reference Product-Test Product (RT) | Fed Cohort: Test Product-Reference Product (TR) | Fed Cohort: Reference Product-Test Product (RT) | Total
Number analyzed (Participants) | 17 | 17 | 25 | 25 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 25 | 25 | 84
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 12 | 6 | 27
  Male | 13 | 12 | 13 | 19 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 17 | 17 | 25 | 25 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 17 | 16 | 24 | 25 | 82
  Other | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Last Observed Concentration at Time t (AUC[0-t]) for Ibuprofen in Fasted Conditions
Description: AUC(0-t) was defined as area under the plasma concentration-time curve from time zero to last observed concentration at time t calculated using the linear up log down trapezoidal rule. Blood samples were collected at indicated timepoints for the analysis of AUC(0-t). Pharmacokinetic (PK) parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose (within 2 hours prior to dosing) and at 5, 10, 15, 20, 30, 45, 60, 75, 90, 105, 120 minutes, 2.5, 3, 4, 6, 8, and 12 hours post-dose
Population: Pharmacokinetic Parameter Set was defined as the evaluable PK parameter data set obtained from randomized participants who received at least one dose of investigational product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter
Groups:
- Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test): Participants received one sachet of ibuprofen arginine granules 400 mg (test product), orally, once on Day 1 of Period 1 or Period 2 as per randomization schedule under fasting conditions. Participants were instructed to take the study product after an overnight fast of at least 10 hours by dissolving it in 240 mL of warm water.
- Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference): Participants received one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 1 or Period 2 as per randomization schedule under fasting conditions. Participants were instructed to take the study product after an overnight fast of at least 10 hours by dissolving it in 240 mL of warm water.
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
hour*micrograms per milliliter | 122.2406 (20.2) | 122.1489 (21.3)
Statistical Analysis 1: Comparison: Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) vs Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference); Test type: Equivalence — The two products were considered to be bioequivalent if 90 percent (%) confidence intervals (CIs) for the geometric mean ratio (GMR) (Test/Reference) for AUC(0-t) were contained within the acceptance interval of 0.8 to 1.25; Geometric Mean Ratio = 1.0008, 90% CI 2-sided [0.9698 to 1.0327]

2. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Time Infinity (AUC [0-inf]) for Ibuprofen in Fasted Conditions
Description: AUC (0-inf) was defined as area under the plasma concentration versus time curve calculated from time 0 to infinity, computed as AUC(0-inf) = AUC(0-t) +Ct/λz where Ct was the plasma concentration at the last measurable sampling time point and λz was the terminal elimination rate constant. Blood samples were collected at indicated timepoints for the analysis of AUC(0-inf). PK parameters were determined by non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
hour*micrograms per milliliter | 124.8000 (21.0) | 124.5173 (22.0)
Statistical Analysis 1: Comparison: Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) vs Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference); Test type: Equivalence — The two products were considered to be bioequivalent if 90% CIs for the GMR (Test/Reference) for AUC (0-inf) were contained within the acceptance interval of 0.8 to 1.25; Geometric Mean Ratio = 1.0023, 90% CI 2-sided [0.9710 to 1.0346]

3. Primary Outcome: Observed Maximum Plasma Concentration (Cmax) for Ibuprofen in Fasted Conditions
Description: Cmax was defined as maximum observed post-dose plasma concentration for ibuprofen. Blood samples were collected at indicated timepoints for the analysis of Cmax. PK parameters were determined by non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
micrograms per milliliter | 54.400 (16.7) | 55.368 (15.9)
Statistical Analysis 1: Comparison: Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) vs Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference); Test type: Equivalence — The two products were considered to be bioequivalent if 90% CIs for the GMR (Test/Reference) for Cmax were contained within the acceptance interval of 0.8 to 1.25; Geometric Mean Ratio = 0.9825, 90% CI 2-sided [0.9383 to 1.0288]

4. Primary Outcome: AUC(0-t) for Ibuprofen in Fed Conditions
Description: AUC(0-t) was defined as area under the plasma concentration-time curve from time zero to last observed concentration at time t calculated using the linear up log down trapezoidal rule. Blood samples were collected at indicated timepoints for the analysis of AUC(0-t). PK parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose (within 2 hours prior to dosing) and 10, 30, 45, 60, 75, 90, 120 minutes, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10 and 12 hours post-dose
Population: Pharmacokinetic Parameter Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter
Groups:
- Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test): Participants received one sachet of ibuprofen arginine granules 400 mg (test product), orally, once on Day 1 of Period 1 or Period 2 as per randomization schedule under fed conditions. Participants were instructed to take the study product after a high-fat/high-calorie meal by dissolving it in 240 mL of warm water.
- Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference): Participants received one sachet of ibuprofen arginine granules 400 mg (Spedifen) (reference product), orally, once on Day 1 of Period 1 or Period 2 as per randomization schedule under fed conditions. Participants were instructed to take the study product after a high-fat/high-calorie meal by dissolving it in 240 mL of warm water.
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 50 | 50
hour*micrograms per milliliter | 114.2490 (18.1) | 115.2125 (18.0)
Statistical Analysis 1: Comparison: Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) vs Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference); Test type: Equivalence — The two products were considered to be bioequivalent if 90% CIs for the GMR (Test/Reference) for AUC(0-t) were contained within the acceptance interval of 0.8 to 1.25; Geometric Mean Ratio = 0.9916, 90% CI 2-sided [0.9755 to 1.0081]

5. Primary Outcome: AUC (0-inf) for Ibuprofen in Fed Conditions
Description: as for outcome 2
Time Frame: as for outcome 4
Population: Pharmacokinetic Parameter Set. Here, overall number analyzed is defined as the number of participants with data available for analysis of this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 44 | 45
hour*micrograms per milliliter | 125.0559 (18.9) | 128.9471 (22.8)
Statistical Analysis 1: Comparison: Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) vs Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 0.9776, 90% CI 2-sided [0.9432 to 1.0133]

6. Primary Outcome: Cmax for Ibuprofen in Fed Conditions
Description: as for outcome 3
Time Frame: as for outcome 4
Population: Pharmacokinetic Parameter Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 50 | 50
micrograms per milliliter | 17.8260 (26.8) | 17.8573 (25.9)
Statistical Analysis 1: Comparison: Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) vs Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference); Test type: Equivalence — The two products were considered to be bioequivalent if 90% CIs for the GMR (Test/Reference) for Cmax were contained within the interval of 0.8 to 1.25; Geometric Mean Ratio = 0.9982, 90% CI 2-sided [0.9431 to 1.0567]

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ibuprofen in Fasted Conditions
Description: Blood samples were collected at indicated timepoints for the analysis of Tmax. PK parameters were determined by non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Set.
Measure: Median (Full Range); unit: hour
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
hour | 0.330 [0.17 to 0.75] | 0.330 [0.17 to 0.50]

8. Secondary Outcome: Elimination Half-life (t1/2) of Ibuprofen in Fasted Conditions
Description: t1/2 was defined as elimination half-life calculated as t1/2 = ln (2)/λz where λz was terminal elimination rate constant. Blood samples were collected at indicated timepoints for the analysis of t1/2. PK parameters were determined by non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter set.
Measure: Median (Full Range); unit: hour
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
hour | 2.2023 [1.7452 to 3.0346] | 2.1300 [1.6851 to 2.7077]

9. Secondary Outcome: Terminal Elimination Rate Constant (λz) of Ibuprofen in Fasted Conditions
Description: λz was defined as terminal elimination rate constant estimated by log-linear regression of the terminal part of the plasma concentration versus time curve. Blood samples were collected at indicated timepoints for the analysis of λz. PK parameters were determined by non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
per hour | 0.3155 (12.8) | 0.3212 (11.9)

10. Secondary Outcome: Percentage of Extrapolated Area of AUC(0-inf) (%AUCex) of Ibuprofen in Fasted Conditions
Description: %AUCex was calculated as %AUCex = (1- AUC[0-t] /AUC[0-inf])*100%. Blood samples were collected at indicated timepoints for the analysis of %AUCex. PK parameters were determined by non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 34 | 34
percentage of AUC | 1.8299 (46.6) | 1.7393 (43.8)

11. Secondary Outcome: Tmax of Ibuprofen in Fed Conditions
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic Parameter Set.
Measure: Median (Full Range); unit: hour
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 50 | 50
hour | 4.500 [0.17 to 10.00] | 4.500 [0.50 to 10.00]

12. Secondary Outcome: t1/2 of Ibuprofen in Fed Conditions
Description: as for outcome 8
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 44 | 45
hour | 2.4053 [1.7676 to 4.6010] | 2.3995 [1.7355 to 10.7675]

13. Secondary Outcome: λz of Ibuprofen in Fed Conditions
Description: as for outcome 9
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 44 | 45
per hour | 0.2653 (27.0) | 0.2515 (39.3)

14. Secondary Outcome: %AUCex of Ibuprofen in Fed Conditions
Description: as for outcome 10
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
Number analyzed (Participants) | 44 | 45
percentage of AUC | 7.9436 (69.8) | 8.3506 (75.4)

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 30 days after the last administration of the investigational product (Up to 42 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) is a particular category of an AE where the adverse outcome is serious. AEs were presented treatment wise.
Arm/Group | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 6/34 | 5/34 | 11/50 | 10/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Test) (N=34) | Fasted Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference) (N=34) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Test) (N=50) | Fed Cohort: Ibuprofen Arginine Granules 400 mg (Spedifen) (Reference) (N=50)
White blood cells urine positive (Investigations) | 3 | 1 | 2 | 2
Blood pressure decreased (Investigations) | 1 | 1 | 5 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 2 | 0
Eosinophil percentage increased (Investigations) | 1 | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3
Urinary occult blood positive (Investigations) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT05737069/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT05737069/SAP_001.pdf